CLINICAL TRIAL: NCT03722147
Title: A Single-arm, Multicenter, Open-label, Phase I/II Study of AK105 as Monotherapy in Relapsed or Refractory Classic Hodgkin Lymphoma
Brief Title: A Study of Anti-PD-1 AK105 in Patients With Relapsed or Refractory Classic Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-201
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hodgkin's Lymphoma
Keywords: immunotherapy; immuno-oncology; Classic Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK105 (Experimental): AK105 200 mg intravenously (IV) every-2-weeks (Q2W)
  Interventions: Biological: AK105

INTERVENTIONS:
Biological: AK105 — AK105 200 mg intravenously (IV) every-2-weeks (Q2W)

SUMMARY:
This is a single-arm, open-label, multicenter, phase I/II study to evaluate efficacy and safety of AK105 in patients with relapsed or refractory classic Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
3. Histologically confirmed classic Hodgkin's lymphoma (cHL) (based on tumor tissue obtained within 3 years prior to enrollment).
4. Relapsed (disease progression during or after most recent therapy) or refractory (failure to achieve CR or PR after most recent therapy) cHL and meet any of the following criterions:

   1. Recurrence or disease progression after autologous hematopoietic stem cell transplantation.
   2. For subject without receiving , the subject has received at least 2 lines of prior systemic chemotherapy. Refractory subject is defined as subject who has not achieved PR after at least 2 cycles of treatment, or subject who has not achieved CR after at least 4 cycles of treatment. If the best response to treatment is PD or the reason for ending the treatment is PD, the subject is consider as refractory without requirement on the number of cycles of treatment that the subject has received. For relapsed subjects, disease progression occurred for the subject who has received at least 2 line of prior systemic chemotherapy.
5. Subject must have at least one measurable lesion (> 1.5 cm in the longest diameter, or > 1 cm in the longest diameter with uptake on 18FDG-PET)according to the Lugano 2014 criteria.
6. Adequate organ functions.
7. Use effective methods of contraception.

Exclusion Criteria:

1. Known nodular lymphoma predominant Hodgkin lymphoma or Grey zone lymphoma.
2. Lymphoma involving the central nervous system.
3. Participated in other clinical studies of experimental drugs or received research treatment or used experimental equipment within 4 weeks prior to the first dose of AK105.
4. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
5. Receipt of the last radiotherapy or the last dose of anticancer therapy (chemotherapy, target therapy, immunotherapy or tumor embolism, etc.) with 4 weeks prior to the first dose of AK105. Receipt of the last dose of nitrocarbamide or mitomycin C within 6 weeks prior to the first dose of AK105.
6. Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTL4 antibody or any other antibody or drug targeting T-cell costimulation or checkpoint pathways such as ICOS, or agonists such as CD40, CD137, GITR, OX40 etc..
7. Had other active malignancies within 5 years prior to enrollment. Locally curable cancer (manifested as cured) is excluded, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
8. Active, known or suspected autoimmune diseases, or a history of the disease within the past 2 years, except the following: vitiligo, alopecia, Graves' disease, psoriasis or eczema that do not require systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring a stable dose of hormone replacement therapy, type I diabetes requiring only a stable dose of insulin replacement therapy, or diseases not expected to recur in the absence of external triggering factors.
9. Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis or chronic diarrhea).
10. Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
11. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
12. History of primary immunodeficiency.
13. History of active tuberculosis.
14. History of allogeneic stem cell transplantation or organ transplantation.
15. Autologous hematopoietic stem cell transplantation performed within 90 days prior to the first dose of AK105.
16. History of gastrointestinal perforation and /or within 6 months prior to enrollment.
17. History of interstitial lung disease.
18. Patients with untreated chronic hepatitis B or with HBV DNA exceeding 500 IU/mL, or with active hepatitis C should be excluded. Inactive HBsAg carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL), or cured hepatitis C patients can be enrolled. For patients with positive HCV antibody, they are eligible to participate in the study only if the test result of HCV RNA is negative.
19. Major surgical procedure (as defined by the investigator) within 30 days prior to the first dose of AK105 or still recovering from prior surgery. Local procedures (eg, placement of a systemic port, core needle biopsy, and prostate biopsy) are allowed if completed at least 24 hours prior to the administration of the first dose of study treatment.
20. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
21. Active infections requiring systemic treatment.
22. Uncontrolled concurrent disease, including but not limited to, persistent or active infection, symptomatic congestive heart failure (according to the New York heart association functional class defined 3 or 4), out of control of high blood pressure, unstable angina, arrhythmia, severe peptic ulcer or gastritis, activity, or mental illness/social status which will limit the participants compliance requirements or damage to the participants to provide written informed consent.
23. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE) (NCI CTCAE v4.03) Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the study drug may be included (eg, hearing loss) after consultation with the medical monitor. Subjects with ≤ Grade 2 neuropathy will be evaluated on a case-by-case basis after consultation with the medical monitor.
24. Receipt of live or attenuated vaccination within 30 days prior to the first dose of AK105, or plan to have live or attenuated vaccination during the study.
25. Known allergy or reaction to any component of the AK105 formulation.
26. History of severe allergic reaction to any other monoclonal antibodies.
27. Women who are pregnant or nursing.
28. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by Independent Radiology Review Committee (IRRC) per the Lugano 2014 Classification | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR, assessed by IRRC per the Lugano 2014 Classification.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of AK105
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
ORR assessed by Investigator | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR, assessed by Investigator per the Lugano 2014 Classification.
Duration of Response (DoR) | Up to 2 years
  From the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to 2 years
  From the first dose of AK105 to the date of the date of objective disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  DCR defined as the proportion of subjects response of CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) per the Lugano 2014 Classification.
Minimum observed concentration (Cmin) of AK105 at steady state | From first dose of AK105 through 30 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through to 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beiing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116